CLINICAL TRIAL: NCT06576713
Title: Identification of the Missing Genetic Causes of Parkinsonian Syndromes: a Combined Approach by Genome and RNA Sequencing
Brief Title: Combined Genome and RNA Sequencing for Genetic Diagnosis of Parkinsonism
Acronym: ParkOmic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9320
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Base Sequence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genome and RNA sequencing (Experimental)
  Interventions: Diagnostic Test: Combiner whole genome and RNA sequencing

INTERVENTIONS:
Diagnostic Test: Combiner whole genome and RNA sequencing — High-throughput DNA and RNA sequencing

SUMMARY:
Despite the increasing availability and advances in the analysis of high-throughput DNA sequencing, the majority of patients with early-onset or familial parkinsonism remain without a molecular diagnosis.

Studying the genetic forms of parkinsonian syndromes presents numerous clinical, scientific and therapeutic interests. In clinical practice, identifying the genetic cause in a patient allow to provide genetic counseling and estimate the risk of recurrence in their relatives. Establishing correlations between the genotype and phenotype of patients with genetically determined parkinsonism, allow to better anticipate the evolution of the disease, or even to highlight biomarkers during the presymptomatic phases. Finally, the proteins encoded by the genes implicated in familial parkinsonism represent potential therapeutic targets likely to be modulated by neuroprotective pharmacological agents, even in sporadic Parkinson's disease.

In this work,investigators aimed at elucidating the missing genetic causes of parkinsonism through the application of combined RNA and whole genome sequencing.

DETAILED DESCRIPTION:
Investigators selected 14 patients with early-onset parkinsonism for whom no variant of certain pathogenicity had been identified after exome sequencing.

Patients and their relatives will have a blood sample collection following the inclusion visit for DNA extraction, patients will receive a skin biopsy for fibroblast culture and RNA extraction for RNA sequencing. The genome sequencing will be performed on an Illumina® HiSeq4000 sequencer.

Investigators will also perform skin biopsies on patients for fibroblast cultures in order to extract RNA for RNA sequencing. The choice of fibroblast analysis for the study of the transcriptome is justified by the fact that genes expressed in the brain likely to be associated with neurodegenerative diseases are more frequently expressed in the skin than in the other clinically accessible tissues such as blood. Skin biopsies will be performed by the referring clinicians, and RNA extraction will be carried out using the Quiagen® RNeasy kit.

Transcriptome analysis by RNA sequencing including sequencing and bioinformatics processing of data, including detection of aberrant splicing (LeafCutter), aberrant expressions (DESeq) and identification of variants (GATK + Varank) will also be carried out Genome data will be integrated with data from RNA sequencing. Investigators plan to analyze all 14 patients according to this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Extrapyramidal syndrome beginning before or at the age of 40 or associated with a family history:
* Dopaminergic denervation proven by ioflupane brain scintigraphy (DaTscan®)
* DNAs from both asymptomatic parents available in biobank
* Subject affiliated to a social protection health insurance scheme or beneficiary or beneficiary
* Subject able to understand the objectives and risks related to the research and to give dated and signed informed consent

Exclusion Criteria:

* - Contraindication for performing a superficial skin biopsy provided for by the protocol
* Molecular cause of parkinsonism previously identified
* Absence of prior genetic exploration by high-throughput DNA sequencing
* Patient with late-onset sporadic parkinsonian syndrome (> 40 years) without family history
* Patient with Parkinson's syndrome associated with a specific diagnosis (genetic or non-genetic pathology: exposure to neuroleptics, toxic origin)
* Impossibility of providing the subject with informed information
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetic diagnosis rate | 18 months
  To estimate the rate of genetic diagnoses obtained by genome sequencing coupled with RNA sequencing within a cohort of patients presenting with early onset or familial parkinsonian syndromes without molecular diagnosis.

SECONDARY OUTCOMES:
Genes implicated | 18 months
  Estimate the proportion of patients carrying pathogenic or probably pathogenic variants in each of the genes identified in this work
Contribution of RNA sequencing | 18 months
  Estimate the proportion of pathogenic or probably pathogenic variants detected secondarily thanks to the contribution of RNA sequencing and not identified by analysis of the genome taken in isolation.
Genotype and Phenotype correlation | 18 months
  Estimate the proportion of patients presenting specific clinical, biological and imaging characteristics for each identified genetic cause (genotype/phenotype correlation).
New genetic causes | 18 months
  Describe new molecular mechanisms of parkinsonian syndromes.
Tolerance | 18 months
  Estimate the proportion of patients experiencing an adverse event related to the procedure.
New associated genes | 18 months
  Describe new genes associated with parkinsonian syndromes.